CLINICAL TRIAL: NCT01013584
Title: The Effect of Weight on Vitamin D Dose Response
Acronym: Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Creighton 8
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Obesity; Vitamin D Deficiency
Keywords: vitamin D
MeSH Terms: conditions — Obesity; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1,000 IU (Active Comparator): 1,000 IU/day of vitamin D3
  Interventions: Dietary Supplement: cholecalciferol
- 5,000 IU (Active Comparator): 5,000 IU/day of vitamin D3
  Interventions: Dietary Supplement: cholecalciferol
- 10,000 IU (Active Comparator): 10,000 IU/day of vitamin D3
  Interventions: Dietary Supplement: cholecalciferol

INTERVENTIONS:
Dietary Supplement: cholecalciferol — daily dose

SUMMARY:
Vitamin D3 is a vitamin that is an essential component of biological regulating systems in humans. Sun exposure is the predominant source of vitamin D3. Previous research has shown that vitamin D3 deficiency is common worldwide. It is especially common in northern countries with long winters due to inadequate sun exposure during winter. In the US, an estimated 36% to 57% of healthy middle-aged to elderly adults have vitamin D3 deficiency. Current research indicates that obesity is associated with a low vitamin D3 level.

DETAILED DESCRIPTION:
Obesity is a known risk factor for vitamin D deficiency. Adequate levels of vitamin D are important, not only for bone health, but appear to be important for prevention of certain autoimmune diseases, infections and cancers. Current FDA recommendations for vitamin D intake do not differentiate between lean and obese people. There are no published studies indicating if the 25(OH)D response to a given daily dose of vitamin D is any less in an obese person than a normal weight person. The purpose of this study is to characterize the quantitative relationship between steady state cholecalciferol input and the resulting serum 25 (OH)D concentration in obese subjects. Data obtained in this study will be compared to published normative data for non-obese subjects. Recommendations will be provided for optimal treatment of vitamin D deficiency in obese men and women.

ELIGIBILITY:
Inclusion Criteria:

* men aged 19 to 60 with BMI > 30.0.
* They will have low (<1,000 IU) usual intake of vitamin D (from milk, multivitamins, supplements, and fortified foods)

Exclusion Criteria:

* Subjects will not have history of hepatic or renal disease.
* Subjects will not be taking medications known to affect vitamin D metabolism such as anti-seizure medications and/or corticosteroids.
* They will not be on hydrochlorothiazide medications which could cause hypercalcemia.
* They will not have diseases causing malabsorption of vitamin D, such as celiac sprue or small bowel surgeries.
* Pregnancy is also an exclusion criterion.

Ages: 19 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2009-11; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To characterize the dose response of 25(OH)D to 1,000, 5,000 or 10,000 IU/day of vitamin D3 for 21 weeks in a group of obese men and women. | 21 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andjela Drincic, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States